CLINICAL TRIAL: NCT05909280
Title: Real-time Pressure Volume Loop Monitoring as a Guide for Enhanced Understanding of Changes in Elemental Cardiovascular Physiology During Therapeutic Strategies Aiming for Hemodynamic Optimization. Cohort I: Veno-arterial Extracorporeal Membrane Oxygenation (PLUTO-I)
Acronym: PLUTO-I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Head of Interventional Cardiology, Principal Investigator, Clinical Professor, Erasmus Medical Center
Other Study IDs: PLUTO-I
Record Dates: First submitted 2023-02-13; First posted 2023-06-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Extracorporeal Membrane Oxygenation; Cardio/Pulm: Heart Failure
Keywords: Pressure-volume loop; Cardiac mechanoenergetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational arm: Patients on VA-ECMO, eligible for weaning
  Interventions: Other: Pressure-volume loop measurements

INTERVENTIONS:
Other: Pressure-volume loop measurements — Pressure-volume loop measurements using a conductance catheter

SUMMARY:
Invasive pressure-volume (PV) loop measurements have the potential to confirm or refute earlier computer simulations and animal studies regarding changes in cardiovascular physiology induced by (veno-arterial) ECMO. PV loop analysis could create a framework for the (ICU-) clinician for VA-ECMO weaning guidance, based on a patient's individual hemodynamic profile. PV loop measurements may, in future, serve as a guide for which patient would benefit most from (prolonged) VA-ECMO support or which patient would require additional LV unloading. Within the context of PLUTO-I, patients on VA-ECMO support who are eligible for weaning from VA-ECMO will undergo biventricular PV loop measurements on different intensities of extracorporeal support.

DETAILED DESCRIPTION:
Using VA-ECMO support, physiological stability can be maintained in patients with refractory hemodynamic failure as bridge to recovery, definitive therapy or decision making. Previous animal studies and computer simulations hypothesize increased LV afterload as well as RV distention during VA-ECMO. Decision making concerning VA-ECMO weaning is largely based on bedside hemodynamic (including echocardiographic) parameters. Profound details of the effects of VA-ECMO on elemental cardiac physiology, including myocardial metabolic efficiency and ventricular-arterial coupling, are limited. We hypothesize biventricular pressure-volume loop (PVL) measurement will enhance understanding of elemental cardiovascular physiology including ventricular interdependence during different levels of VA-ECMO support. PVL measurement will hypothetically provide opportunities in discovering novel predictors for successful weaning from VA-ECMO support. For the purpose of PLUTO-I, patients on VA-ECMO who are eligible to wean will undergo invasive PV-loop measurements on different intensities of extracorporeal flow.

ELIGIBILITY:
Inclusion Criteria:

- On VA-ECMO support for any indication

Exclusion Criteria:

* Age < 18 years
* Re-initiation of VA-ECMO during the same ICU admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients on VA-ECMO support for any indication
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Stroke Work in mmHg/mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  The energy necessary for the myocardium to propel blood in the ventricle. Expressed by PV-loop reconstructions based on conductance catheter measurements.
Potential Energy in mmHg/mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  The (unused) energy stored in the myocardium following systole. Expressed by PV-loop reconstructions based on conductance catheter measurements.
Pressure-Volume Area in mmHg/mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  The net metabolic demand of the myocardium throughout the cardiac cycle. Expressed by PV-loop reconstructions based on conductance catheter measurements.

SECONDARY OUTCOMES:
Stroke Volume in mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements.
Cardiac Output | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  By thermodilution, using pulmonary artery catheterization
Preload recruitable stroke work in mmHg/mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements.
Tau in ms | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements.
Systolic and diastolic intraventricular dyssynchrony in % | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements.
Minimal and maximal dP/dt in mmHg/s | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements.
Arterial elastance (Ea) and end-systolic elastance (Ees) in mmHg/mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements (following application of concerning single-beat algorithms)
End-diastolic and end-systolic pressure in mmHg | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements.
End-diastolic and end-systolic volume in mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements.
Starling Contractile Index in mmHg/mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  Expressed by PV-loop reconstructions based on conductance catheter measurements.
V0, V15, V30 and V100 in mL | Perprocedural (i.e. when ECMO flow is decreased from maximal to minimal L/min)
  I.e. ventricular volume at 0, 15, 30 and 100 mmHg, expressed by PV-loop reconstructions based on conductance catheter measurements.
All-cause mortality | Within 30 days after study measurements
  Mortality, irrespective of etiology
Successful weaning from VA-ECMO | 48 hours after study measurements
  A state of persistent hemodynamic stability without the necessity for re-initiation of VA-ECMO support within 48 hours after termination of VA-ECMO support as well as survival at least 48 hours after decannulation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Van Mieghem, Prof MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No